CLINICAL TRIAL: NCT05510960
Title: Video Gaming Improves Robotic Surgery Simulator Success: A Multi-clinic Cross-sectional Study on Robotic Skills
Brief Title: Video Gaming Improves Robotic Surgery Simulator Success
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mustafa Özgür Kılınçarslan, Principal investigator, Ege University
Other Study IDs: 21-3T/17
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Robotic Surgery; Simulator
Keywords: robotic surgery; simulation-based learning; video game experience; surgical education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General surgery residents: 39 participants
  Interventions: Other: Video game & Robotic surgery simulator success
- Urology residents: 14 participants
  Interventions: Other: Video game & Robotic surgery simulator success
- Pediatric surgery residents: 7 participants
  Interventions: Other: Video game & Robotic surgery simulator success

INTERVENTIONS:
Other: Video game & Robotic surgery simulator success — A questionnaire was administered to all participants, asking about their demographic information, surgical experience, hobbies, and previous video game playing experiences.
  After the questionnaire, the participants were asked to play the Temple Run (Imangi Studios, NC, USA) and Piano Tiles 2™ mobile games for one month. At the end of the period, with the da Vinci® Skills Simulator™ for one hour, all participants performed four different robotic surgery simulator tasks (Camera Targeting 1, Energy Switching 1, Ring & Rail 2, Vertical Defect Suturing) that require the ability to apply basic robotic surgery rules and measure surgical skills.

SUMMARY:
Investigators aimed to investigate the effects of video game habits, duration of experience, and training in different surgical clinics on the success of robotic surgery simulators.

In this prospective, observational, comparative, and multi-clinic study, all participants played the Temple Run and Piano Tiles 2™ mobile games for one month after responding to a questionnaire including their sociodemographic characteristics, surgical experience, and past and current video game experience. At the end of the study period, participants experienced four different robotic surgery simulator tasks (Camera Targeting 1, Energy Switching 1, Ring & Rail 2, Vertical Defect Suturing) in the da Vinci® Skills Simulator™. Additionally, sociodemographic data were statistically analyzed with mobile game scores, and 13 different performance scores were obtained from the simulator.

ELIGIBILITY:
Inclusion Criteria:

* To be a physician trained in Surgery in the Department of General Surgery. Pediatric Surgery and Urology.
* To be an assistant and specialist of the departments with robotic surgery experience.
* To be acquainted with laparoscopic surgery.
* Having played video games.

Exclusion Criteria:

* Participation in our study is on a voluntary basis and we have no criteria other than physicians who want to leave the study voluntarily.

Ages: 24 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents from general surgery, urology, and pediatric surgery clinics were included in the study. Sixty of the 64 total participants completed all the processes. Four participants were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Robotic surgery simulator score of participants by video game experience | 2 months
  The effect of both previous and current video game on simulator results

SECONDARY OUTCOMES:
Determination of robotic surgery success among clinics according to simulator score | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data of participants will be kept confidential.

REFERENCES:
- [Derived] Kilincarslan O, Turk Y, Vargor A, Ozdemir M, Hassoy H, Makay O. Video gaming improves robotic surgery simulator success: a multi-clinic study on robotic skills. J Robot Surg. 2023 Aug;17(4):1435-1442. doi: 10.1007/s11701-023-01540-y. Epub 2023 Feb 8. PMID 36754922